CLINICAL TRIAL: NCT02529371
Title: Pre-Marketing Feasibility Evaluation of the UriCap-RM - Urine Collection in Hospitalized Male Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: G.R. Dome Medical Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: GRD-01M
Record Dates: First submitted 2015-08-16; First posted 2015-08-20 (Estimated); Last update posted 2015-09-18 (Estimated); Status verified 2015-09

CONDITIONS: Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- UriCap-RM (Experimental): The device is comprised of a reusable part and a single use adhesive tape. The device is removed once daily and the reusable part is rinsed, dried and reapplied with a new adhesive tape.
  Interventions: Device: UriCap-RM

INTERVENTIONS:
Device: UriCap-RM — UriCap-RM is comprised of a reusable part and a single use adhesive tape. The reusable part is applied over the urethral meatus and is held in position by a stabilizer and adhesive tape. It is connected to a standard urine collection bag. The UriCap-RM is used on male patients who would otherwise use diapers, a condom-type urine collection device or an indwelling catheter for urine collection.
  Other Names: non-invasive urine collection device

SUMMARY:
The study will evaluate device performance and user satisfaction in the UriCap-RM, an FDA cleared non-invasive urine collection device for men.

DETAILED DESCRIPTION:
Following various disease conditions such as trauma, orthopedic surgery, and infections etc., patients may be bedridden and unable to void in a bedpan or to make their way to the toilet. Others may be incontinent of urine. In such situations an indwelling catheter is often placed to relieve patients while they are incapacitated; in many cases a catheter is placed despite lack of urinary retention. Indwelling catheters, although effective, are associated with discomfort, pain, and urinary tract infections. In other cases diapers or absorbent pads may be used, or a condom-type urine collection device. These may be associated with skin irritation and infection.

The study will evaluate the UriCap-RM non-invasive urine collection device in hospitalized men.

ELIGIBILITY:
Inclusion Criteria:

* Male ≥ 18 years old.
* Empties the bladder completely on voiding
* A clinical indication for an indwelling catheter, use of pads or diapers
* Subject has signed an informed consent form, is cooperative and willing to complete all study procedures
* Absence of localized disease at the site of device application - no discharge, itching, inflammation or skin condition - - on visual examination
* Subject has no hypersensitivity to silicon.

Exclusion Criteria:

* Known allergy to silicon
* Dysuria
* Urinary retention - Post-void residual urine more than 300cc
* Hematuria or pyuria (turbidity) on visual inspection, according to investigator judgement.
* Diagnosed with acute renal failure, according to investigator judgement.
* Serious or unstable psychological condition (e.g., eating disorders, clinical depression, anxiety, emotionally labile) which, in the opinion of the Investigator, would compromise the subject's well-being or successful participation in the study
* Participating in another clinical study.
* Financial interest in the Sponsor Company or a competitor company by subject or a family member

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2015-09; Primary Completion 2015-10 (Estimated); Study Completion 2015-10 (Estimated)

PRIMARY OUTCOMES:
Performance of the device in collecting urine | 1-30 days
  Multiple variables will be assessed and their measurements aggregated to arrive at number of events reported:
  * Patient's anatomy does not enable application of the device
  * Leakage
  * Pooling of urine in the tubing
  * Tubing disconnections
  * Adhesive tape disconnections
  * Need for repositioning of device
  * Device malfunctions
Patient Comfort | 1-30 days
  Daily assessment of comfort rated in the "Universal Pain Assessment Scale" of 1-10.
Healthcare provider (HCP) satisfaction in device use | up to 60 days
  Nurses will fill a "Treatment Satisfaction Questionnaire" once after termination of all study patients
Patient Satisfaction in Device Use | 1-30 days
  Administration of a "Treatment Satisfaction Questionnaire" at termination of device use.

SECONDARY OUTCOMES:
Effectiveness of defined device cleaning procedure | 1-30 days
  The reusable part will be visually inspected after cleaning for suitability for reuse. Devices which exhibit any of the following properties will be discarded: color change, residual soiling, loss of mechanical integrity, torn, rough edges. The effectiveness of the cleaning procedure will be measured as the average number of days the device can be reused.
Number of leakage events resulting from device movement | 1-30 days
Number of patients with Adverse Events that are related to device use | 1-30 days

CONTACTS AND LOCATIONS:
Overall Officials: Elad Schiff, MD, Principal Investigator — no affiliation